CLINICAL TRIAL: NCT00003548
Title: Phase I Study of Intraperitoneal Administration of 9-Amino-20(S)-Camptothecin to Patients With Cancer Predominantly Confined to the Peritoneal Cavity
Brief Title: Aminocamptothecin in Treating Patients With Advanced Cancer of the Peritoneal Cavity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066605; U01CA076642 (NIH); P30CA016087 (NIH); NYU-9753; NCI-T97-0123
Record Dates: First submitted 2000-05-02; First posted 2004-02-20 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Cancer
Keywords: stage IV colon cancer; stage IV breast cancer; recurrent breast cancer; stage IV gastric cancer; recurrent gastric cancer; recurrent pancreatic cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; stage IV anal cancer; recurrent anal cancer; stage IV esophageal cancer; recurrent esophageal cancer; stage IV cervical cancer; recurrent cervical cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; stage IV vulvar cancer; recurrent vulvar cancer; stage IVA vaginal cancer; stage IVB vaginal cancer; recurrent vaginal cancer; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; advanced adult primary liver cancer; recurrent adult primary liver cancer; recurrent gestational trophoblastic tumor; stage IV endometrial carcinoma; recurrent endometrial carcinoma; unresectable gallbladder cancer; recurrent gallbladder cancer; unresectable extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; recurrent small intestine cancer; carcinoma of the appendix; fallopian tube cancer; stage IV uterine sarcoma; recurrent uterine sarcoma; recurrent carcinoma of unknown primary; stage IV pancreatic cancer
MeSH Terms: conditions — Neoplasms; Colonic Neoplasms; Breast Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms; Rectal Neoplasms; Anus Neoplasms; Esophageal Neoplasms; Uterine Cervical Neoplasms; Carcinoma, Ovarian Epithelial; Vulvar Neoplasms; Vaginal Neoplasms; Carcinoma, Hepatocellular; Gestational Trophoblastic Disease; Endometrial Neoplasms; Gallbladder Neoplasms; Bile Duct Neoplasms; Appendiceal Neoplasms; Fallopian Tube Neoplasms; Neoplasms, Unknown Primary

INTERVENTIONS:
Drug: aminocamptothecin colloidal dispersion

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of aminocamptothecin in treating patients with advanced cancer of the peritoneal cavity.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the qualitative and quantitative toxicities of intraperitoneal aminocamptothecin colloidal dispersion administered every 28 days in 6 applications over a 12 day period in patients with advanced cancer confined to the peritoneal cavity. II. Determine the maximum tolerated dose of aminocamptothecin colloidal dispersion on this novel schedule in this patient population. III. Obtain pharmacological and biochemical data as potential predictors of responses and/or drug toxicities in these patients. IV. Document the presence and degree of antitumor activity of this regimen in this patient population.

OUTLINE: This is a dose escalation study. Patients receive intraperitoneal aminocamptothecin colloidal dispersion (9-AC) over 30-60 minutes in 6 applications over a 12 day period (days 1, 3, 5, 8, 10, and 12). Courses are repeated every 28 days. Treatment continues for 4-6 courses in the absence of unacceptable toxic effects or disease progression. The dose of 9-AC is escalated in cohorts of 3-6 patients until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose limiting toxicity. Patients are followed until death.

PROJECTED ACCRUAL: Approximately 15-20 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed advanced malignancy involving the peritoneal cavity, excluding leukemia and lymphoma Patients with ovarian cancer must have received prior standard therapy Predominantly small tumor metastases less than 1.0 cm in diameter including: Ovarian cancer with epithelial histology Other gynecological tumors Breast cancer Gastric cancer Colorectal cancer Appendiceal cancer Pancreatic cancer Unknown primary cancer Other malignancies with predominantly intraperitoneal manifestation No extensive intraperitoneal adhesions that cannot be easily lysed laparoscopically or by laparotomy No symptomatic disease outside the peritoneal cavity Asymptomatic disease outside the peritoneum considered (e.g., bone lesions)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 3 months Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2.0 mg/dL AST no greater than 2 times upper limit of normal Renal: Creatinine no greater than 2.0 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas and/or mitomycin) Endocrine therapy: Not specified Radiotherapy: At least 3 weeks since prior radiotherapy Surgery: See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 1998-08; Primary Completion 2001-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco M. Muggia, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States